CLINICAL TRIAL: NCT02173587
Title: Efficacy of Thick Shell Mussel Lipid Extract in Chinese Subjects With Rheumatoid Arthritis
Brief Title: Study Evaluating the Efficacy of Thick Shell Mussel Lipid Extract in Chinese Subjects With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Duo li, Study director, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NNSFC81273064
Record Dates: First submitted 2014-06-22; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Anti-inflammation, Rheumatoid arthritis, Thick shell mussel lipid extract, Chinese
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mussel oil capsules (Experimental): Four mussel oil capsules (containing 800mg mussel oil and 800mg corn oil) per day for first two months and two mussel oil capsules (containing 400mg mussel oil and 400mg corn oil) per day thereafter for four months.
  Interventions: Dietary Supplement: Mussel oil capsules
- Corn oil capsuels (Placebo Comparator): Four corn oil capsules (containing 1600mg corn oil) for first two months and two mussel oil capsules (containing 800mg corn oil) per day thereafter for four months.
  Interventions: Dietary Supplement: Corn oil capsules

INTERVENTIONS:
Dietary Supplement: Mussel oil capsules — Each mussel oil capsule contained 200mg thick shell mussel lipid extract and 200mg corn oil.Each patient in this group received daily four mussel oil capsules (containing 800mg mussel oil and 800mg corn oil) for first two months and two mussel oil capsules per day thereafter
  Other Names: lipid extract from hard-shelled mussel (Mytilus coruscus)
  Arms: Mussel oil capsules
Dietary Supplement: Corn oil capsules — Each corn oil capsule contained 400mg corn oil.Each patient in this group received daily four corn oil capsules (1600mg corn oil) for first two months and two corn oil capsules per day thereafter
  Other Names: Placebo comparator
  Arms: Corn oil capsuels

SUMMARY:
Previous study found that lipid extract from hard-shelled mussel (HMLE) at a dose of 100mg/kg possessed strong anti-inflammatory activity by diminishing the hind paw swelling and arthritis index in rat model. In the present study, HMLE was processed to capsules under strict food safety supervision and patients with active rheumatoid arthritis (RA）were selected to examine whether supplementation with HMLE could improve clinical and laboratory parameters of disease activity. The validated disease activity score that include 28 joint counts and ESR (DAS28) and validated clinical disease activity index (CDAI) were primary outcome measure. Laboratory parameters including IL-1β, IL-6, IL-10, TNF-α,PGE2 and COX-2 were also measured to explore the mechanisms.

DETAILED DESCRIPTION:
In this randomized controlled design, patients continued receiving background medications (slow-acting anti-rheumatic drugs and non-steroidal anti-inflammatory drugs) without change and were assigned to two groups. The first group (G1) received daily four mussel oil capsules (containing 800mg mussel oil and 800mg corn oil) for first two months and two mussel oil capsules per day thereafter. The second group (G2) received corn oil capsules (400mg corn oil per capsule) according to the same regimen. All patients were asked to keep a 7-day food diary before intervention and during wk 12. Dietary energy and nutrient intake of each subject during the preexperimental and study period were assessed from the dietary records by using "Diet Analysis" software (Cao Aihong, Taiyuan, China). All the enrolled patients visited Zhejiang Sir Run Run Shaw Hospital in the morning following an overnight fast at baseline and 3-month intervals, and underwent anthropometric measurements including height, body weight, waist circumference, hip circumference, heart rate and blood pressure. Then clinical evaluations were performed during face-to-face interview by a professional attending doctor and ten milliliter of peripheral venous blood was drawn. Serum and erythrocyte samples were also promptly processed and frozen at -80℃ until analysis.

ELIGIBILITY:
Inclusion Criteria:

* According to the American College of Rheumatology criteria, patients from Zhejiang province with active RA were included in this study and all participants were Chinese. Patients had at least 3 swollen joints and 6 tender joints or had an erythrocyte sedimentation rate (ESR) of >28mm/hr or morning stiffness of at least 45 min were classified as with active disease.

Exclusion Criteria:

* Subjects suffering hyperlipidemia, hyperglycemia, diabetes mellitus, cardiovascular diseases, gastrointestinal problems, liver and renal failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Disease activity score that include 28 joint counts and ESR (DAS28) | Six months (3-month intervals)
  The validated disease activity score that include 28 joint counts and ESR (DAS28) were primary outcome measure. DAS28 was calculated as the formula: DAS28=[0.56*sqrt（T28）+0.28*sqrt（SW28）+0.70*Ln（ESR）]*1.08+0.16.
  T28: Tender joint count; SW28: Swollen joint count; ESR: Erythrocyte sedimentation rate.
  T28 and SW28 were determined by a professional doctor who was blind to the patient groups and ESR (Westergreen's method) was analyzed on Monitor 20 (VITAL Diagnostics, Italy).

OTHER OUTCOMES:
C-reactive protein | 6 months (3-month intervals)
  Fasting blood specimens were obtained from all participants at entry, 12 and 24 wk later. C-reactive protein was analyzed on HITACHI 7020 chemistry analyzer using enzymebased colorimetric test or colorimetric test supplied by DiaSys Diagnostic Systems (Shanghai) Co., Ltd. within four hours of blood collection.
Rheumatoid factor | 6 months (3-month intervals)
  Fasting blood specimens were obtained from all participants at entry, 12 and 24 wk later.Rheumatoid factor were analyzed on HITACHI 7020 chemistry analyzer using enzymebased colorimetric test or colorimetric test supplied by DiaSys Diagnostic Systems (Shanghai) Co., Ltd. within four hours of blood collection.
Prostaglandin E2 (PGE2) | 6 months (3-month intervals)
  Levels of PGE2 from serum were determined by the research workers who were blind to the patient groups using ELISA Kits (Nanjing Jiancheng Technology Co., Lte., Nanjing, China), according to the manufacturer's instructions.
Interleukin-1β(IL-1β) | 6 months (3-month intervals)
  Levels of IL-1β from serum were determined by the research workers who were blind to the patient groups using ELISA Kits (Nanjing Jiancheng Technology Co., Lte., Nanjing, China), according to the manufacturer's instructions.
Tumor necrosis factor-α (TNF-α) | 6 months (3-month intervals)
  Levels of TNF-α from serum were determined by the research workers who were blind to the patient groups using ELISA Kits (Nanjing Jiancheng Technology Co., Lte., Nanjing, China), according to the manufacturer's instructions.
Interleukin-6 (IL-6) | 6 months (3-month intervals)
  Levels of IL-6 from serum were determined by the research workers who were blind to the patient groups using ELISA Kits (Nanjing Jiancheng Technology Co., Lte., Nanjing, China), according to the manufacturer's instructions.
Interleukin-10 (IL-10) | 6 months (3-month intervals)
  Levels IL-10 from serum were determined by the research workers who were blind to the patient groups using ELISA Kits (Nanjing Jiancheng Technology Co., Lte., Nanjing, China), according to the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Duo Li, Dr., Study Director — Department of Food Science and Nutrition, Zhejiang University
Locations (1):
- Zhejiang university, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Fu Y, Li G, Zhang X, Xing G, Hu X, Yang L, Li D. Lipid extract from hard-shelled mussel (Mytilus coruscus) improves clinical conditions of patients with rheumatoid arthritis: a randomized controlled trial. Nutrients. 2015 Jan 16;7(1):625-45. doi: 10.3390/nu7010625. PMID 25602164